CLINICAL TRIAL: NCT02741856
Title: SCOPE2 - A Randomised Phase II/III Trial to Study Radiotherapy Dose Escalation in Patients With Oesophageal Cancer Treated With Definitive Chemo-radiation With an Embedded Phase II Trial for Patients With a Poor Early Response Using Positron Emission Tomography (PET)
Brief Title: Study of Chemoradiotherapy in Oesophageal Cancer Including PET Response and Dose Escalation
Acronym: SCOPE2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lisette Nixon (Other Government)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor-Investigator, Lisette Nixon, Senior Trial Manager, Velindre NHS Trust
Organization: Velindre NHS Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/VCC/0015; 2015-001740-11 (EudraCT Number); Ethics Reference Number (Other: 15/WA/0395)
Record Dates: First submitted 2016-04-12; First posted 2016-04-18 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Carboplatin; Paclitaxel; Cisplatin; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (carboplatin/paclitaxel+standard RT dose) (Experimental): Cycle 1: Week 1-3: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-21
  Cycle 2: Week 4-6: carboplatin AUC 5 on D1 and paclitaxel 175mg/m2 on D1
  Week 7-11: Weekly carboplatin AUC 2 and paclitaxel 50mg/m2 concomitant with radiotherapy (50Gy/25 fractions)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Cisplatin; Drug: Capecitabine; Radiation: Radiotherapy
- Arm 2 (cisplatin/capecitabine+standard RT dose) (Experimental): Cycle 1: Week 1-3: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-21
  Cycle 2: Week 4-6: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-21
  Cycle 3: Week 7-9: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-21
  Cycle 4: Week 10-11: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-14
  Cycles 3 and 4 are given concomitantly with radiotherapy (50Gy/25 fractions). Capecitabine stops on last day of RT.
  Interventions: Drug: Cisplatin; Drug: Capecitabine; Radiation: Radiotherapy
- Arm 3 (carboplatin/paclitaxel+high RT dose) (Experimental): Cycle 1: Week 1-3: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-21
  Cycle 2: Week 4-6: carboplatin AUC 5 on D1 and paclitaxel 175mg/m2 on D1
  Week 7-11: Weekly carboplatin AUC 2 and paclitaxel 50mg/m2 concomitant with radiotherapy (60Gy/25 fractions)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Cisplatin; Drug: Capecitabine; Radiation: Radiotherapy
- Arm 4 (Cisplatin+Capecitabine+high RT dose) (Experimental): Cycle 1: Week 1-3: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-21
  Cycle 2: Week 4-6: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-21
  Cycle 3: Week 7-9: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-21
  Cycle 4: Week 10-11: cisplatin 60mg/m2 on D1 and capecitabine 625mg/m2 bd D1-14 Cycles 3 and 4 are given concomitantly with radiotherapy (60Gy/25 fractions). Capecitabine stops on last day of RT.
  Interventions: Drug: Cisplatin; Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Carboplatin — For more information please see the arm descriptions section.
  Arms: Arm 1 (carboplatin/paclitaxel+standard RT dose); Arm 3 (carboplatin/paclitaxel+high RT dose)
Drug: Paclitaxel — For more information please see the arm descriptions section.
  Arms: Arm 1 (carboplatin/paclitaxel+standard RT dose); Arm 3 (carboplatin/paclitaxel+high RT dose)
Drug: Cisplatin — For more information please see the arm descriptions section.
Drug: Capecitabine — For more information please see the arm descriptions section.
Radiation: Radiotherapy — For more information please see the arm descriptions section.

SUMMARY:
Research has shown that increasing the dose of radiotherapy improves outcomes in patients with lung and head and neck cancers. This study aims to see whether this is also the case for patients with tumour of the oesophagus. This trial will compare the effects of the standard dose of radiotherapy to a higher dose whilst closely monitoring the side effects.

A comparison will also be made regarding the effects of the standard drugs used in chemotherapy (cisplatin and capecitabine) with an alternative combination (carboplatin and paclitaxel) in patients that do not show a response to chemotherapy with standard drugs early on in treatment.

All patients will receive 6 weeks of chemotherapy and 5 weeks of chemoradiotherapy.

How the study will be conducted:

Prior to the commencement of treatment each patient will have a special scan called a PET scan. Patients will receive a second PET scan two weeks after the start of standard chemotherapy. The changes between the two scans will then be used to allocate treatment into the different arms of the study. All study subjects will be randomised to receive either the standard radiotherapy dose or the high radiotherapy dose. The participants that do not respond to the first cycle of standard chemotherapy will be eligible to take part in the aspect of the trial looking at an alternative chemotherapy regimen. Patients will be randomised as follows;

On the basis of the second PET scan, patients who are not responding to standard chemotherapy will be allocated by a computer to one of the four groups detailed below:

* Standard chemotherapy and standard dose of radiotherapy
* Standard chemotherapy and higher dose of radiotherapy
* Alternative chemotherapy and standard dose of radiotherapy
* Alternative chemotherapy and higher dose of radiotherapy

Patients who are responding to standard chemotherapy (or where the response is unknown or those who were not eligible for PET scan portion of the study) will be allocated by a computer to one of two groups detailed below:

* Standard chemotherapy and standard dose of radiotherapy
* Standard chemotherapy and higher dose of radiotherapy

The arms within each of the groups above (responders and non-responders) will be equal in size and patients will be allocated randomly by a computer.

This study will also compare the way that this treatment affects the two different cell types found in oesophageal tumours.

The effects of the different treatment, together with the costs of the different treatment and the effects on quality of life will be analysed to see which is more effective for each of the different groups.

ELIGIBILITY:
Main inclusion criteria:

1. 17 years of age or older.
2. Have been selected to receive potentially curative definitive chemoradiotherapy by a specialist Upper GI MDT.
3. Histologically confirmed adenocarcinoma, undifferentiated cancer or squamous cell carcinoma.
4. Tumours of the cervical, thoracic oesophagus, or gastro-oesophageal junction (GOJ) with proximal extent of disease no more proximal than 15cm ab oral and distal extent of primary tumour no more than 2 cm beyond the GOJ.
5. Tumours staged with endoscopic ultrasound*, CT and PET-CT to be T1-4 and N+/- (provided total tumour length including nodes is ≤10).
6. Total contiguous disease length ≤10cm defined by CT, EUS and/or PET. The primary tumour should also be ≤8cm.
7. WHO performance status 0 or 1.
8. Adequate cardiovascular function for safe delivery of chemo-radiation in the opinion of the principal investigator. Where there is clinical concern patients should have an adequate cardiac ejection fraction ≥ 40% as determined by MUGA scan or ECHO (within 4 weeks prior to enrolment).
9. Adequate respiratory function for safe delivery of chemo-radiation in the opinion of the Principal Investigator. Where there is clinical concern FEV1 ≥ 1 litre as determined by spirometry (within 4 weeks prior to enrolment).
10. Patients with clinically significant hearing impairment (hearing loss with hearing aid, or hearing loss where intervention indicated, or limiting daily activities or tinnitus limiting daily activities or sensory-motor neuropathy are eligible, however, cisplatin will be replaced by carboplatin (AUC 5)
11. Adequate haematological, hepatic and renal function
12. Patients agree to use effective forms of contraception during the trial (if applicable to patient).
13. Patients who have provided written informed consent prior to enrolment.

    Additional inclusion criteria for patient eligibility for PET randomisation (cisplatin/capecitabine vs carboplatin/paclitaxel) as assessed at local centre:
14. Baseline SUVmax ≥ 5.
15. PET scan 14 days after start of chemo (-2/+3 days from this date is acceptable)
16. Not responding to early cis/cape chemotherapy (this is defined as patients having a <35% reduction in SUVmax)

18. To be eligible for PET randomisation, the baseline PET-CT must have been within 4 weeks prior to start date of treatment.

Patients that are eligible for the trial but are ineligible for PET randomisation will be randomised to receive 50/60Gy radiotherapy plus cisplatin and capecitabine.

* Patients where the EUS scope is unable to pass are eligible.

Main exclusion criteria:

1. Patients who have had previous treatment for invasive oesophageal carcinoma or gastro-oesophageal junction carcinoma (not including PDT or laser therapy for high grade dysplasia/carcinoma in-situ).
2. Patients with metastatic disease i.e. M1a or M1b according to UICC TNM version 7.
3. Patients with other active malignancy or past malignancy in remission for less than 3 years are not eligible for the trial. However, patients with the following conditions which have been curatively treated will NOT be excluded: basal cell carcinoma, carcinoma-in-situ breast and carcinoma-in-situ cervix.
4. Patients with >2cm mucosal extension of tumour into the stomach or where the superior extent is proximal to 15 cm ab oral.
5. Patients with unstable angina or uncontrolled hypertension or cardiac failure or other clinically significant cardiac disease.
6. Patients who need continued treatment with a contraindicated concomitant medication or therapy.
7. Patients with known dihydropyrimidine dehydrogenase (DPD) deficiency.

9. Patients with serious infections

10. Known hypersensitivity to IMPs.

11. Women who are pregnant or breastfeeding.

12. Oesophageal stent (patients requiring a PEG/RIG/feeding jejunostomy for nutritional purposes are eligible).

13. Any other situation, which in the opinion of the local PI, makes the patient an unsuitable candidate for this trial.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2016-11-04 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint phase II in squamous cell carcinoma comparing standard dose radiotherapy to high dose radiotherapy | 24 weeks
  24 week treatment failure free survival (TFFS).
Primary endpoint phase III in squamous cell carcinoma: Overall survival (OS) comparing standard dose radiotherapy to high dose radiotherapy | 24 weeks
  Overall survival (OS)
Primary endpoint in squamous cell carcinoma when switching chemotherapy | 24 weeks
  24 week treatment failure free survival (TFFS).
Primary endpoint phase in adenocarcinoma phase II comparing standard dose radiotherapy to high dose radiotherapy | 24 weeks
  24 week treatment failure free survival (TFFS).
Primary endpoint in adenocarcinoma when switching chemotherapy | 24 weeks
  24 week treatment failure free survival (TFFS).

SECONDARY OUTCOMES:
Overall survival | 5 years follow up
  Overall survival assessed at each visit. Additionally patients will be flagged with the HSCIC to reduce loss to follow up.
Progression free survival | 5 years
  Progression free survival (PFS), additionally patients will be flagged with the HSCIC to reduce loss to follow up.
Quality of Life | Baseline, week 7, end of treatment, 6, 12 and 24 months
  Quality of Life (QoL): EORTC QLQ-C30 and EORTC QLQ-OES18 questionnaires
Toxicity | After each treatment cycle and at follow up visits
  CTCAE v4.03 at baseline, after each treatment cycle, and follow up visits. Patients in the dose escalation arm will have additional assessment and 6 and 9 weeks post RT to monitor toxicities.
Health economics | Baseline, end of treatment, 6, 12 and 24 months
  Health economic data will be collected using health resource utilisation log plus data on health resource usage

CONTACTS AND LOCATIONS:
Overall Officials: Tom Crosby, Principal Investigator — Velindre University NHS Trust
Locations (26):
- United Kingdom (26):
  - Aberdeen Royal Infirmary, Aberdeen
  - Bristol Haematology & Oncology, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Kent and Canterbury, Canterbury
  - Velindre Cancer Care Centre, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - University Hospital Coventry, Coventry
  - Derby Teaching Hospitals NHS Trust, Derby
  - Glan Clwyd Hospital, Glan Clwyd
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Gloucestershire Royal Hospital, Gloucester
  - Castle Hill Hospital, Hull
  - The Clatterbridge Cancer Centre nhs Foundation Trust, Liverpool
  - Guy's and St Thomas', London
  - Imperial College Healthcare NHS Trust, London
  - North Middlesex Hospital, London
  - The Royal Marsden Hospitals (Fulham), London
  - The James Cook University Hospital, Middlesbrough
  - Churchill Hospital, Oxford
  - Peterborough and Stamford Hospitals NHS Foundation Trust, Peterborough
  - Sheffield Teaching Hospitals - Weston Park Hospital, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - The Royal Marsden Hospitals (Sutton, Surrey), Sutton
  - Singleton Hospital, Swansea
  - Worcestershire Royal Hospital, Worcester
  - Wrexham Maelor, Wrexham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Holland-Hart D, Longo M, Bridges S, Nixon L, Hawkins M, Crosby T, Nelson A. A qualitative study exploring participants' experiences of the SCOPE2 trial: chemoradiotherapy dose escalation in oesophageal cancer. Trials. 2025 Feb 26;26(1):70. doi: 10.1186/s13063-025-08768-z. PMID 40012034
- [Derived] Holland-Hart D, Longo M, Bridges S, Nixon LS, Hawkins M, Crosby T, Nelson A. The experiences of patients with oesophageal cancer receiving chemoradiotherapy treatment: a qualitative study embedded in the SCOPE2 trial. BMJ Open. 2024 Sep 23;14(9):e076394. doi: 10.1136/bmjopen-2023-076394. PMID 39313288
- [Derived] Mukherjee S, Hurt CN, Adams R, Bateman A, Bradley KM, Bridges S, Falk S, Griffiths G, Gwynne S, Jones CM, Markham PJ, Maughan T, Nixon LS, Radhakrishna G, Roy R, Schoenbuchner S, Sheikh H, Spezi E, Hawkins M, Crosby TDL. Efficacy of early PET-CT directed switch to carboplatin and paclitaxel based definitive chemoradiotherapy in patients with oesophageal cancer who have a poor early response to induction cisplatin and capecitabine in the UK: a multi-centre randomised controlled phase II trial. EClinicalMedicine. 2023 Jun 26;61:102059. doi: 10.1016/j.eclinm.2023.102059. eCollection 2023 Jul. PMID 37409323
- [Derived] Sakanaka K, Ishida Y, Fujii K, Ishihara Y, Nakamura M, Hiraoka M, Mizowaki T. Radiation Dose-escalated Chemoradiotherapy Using Simultaneous Integrated Boost Intensity-Modulated Radiotherapy for Locally Advanced Unresectable Thoracic Oesophageal Squamous Cell Carcinoma: A Single-institution Phase I Study. Clin Oncol (R Coll Radiol). 2021 Mar;33(3):191-201. doi: 10.1016/j.clon.2020.07.012. Epub 2020 Aug 4. PMID 32768158